CLINICAL TRIAL: NCT01880853
Title: Ultrasound and Mammography for Screening Breast Cancer in Chinese Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PUMCH-breast-screening
Record Dates: First submitted 2013-06-14; First posted 2013-06-19 (Estimated); Last update posted 2013-09-10 (Estimated); Status verified 2013-09

CONDITIONS: Breast Cancer
Keywords: breast cancer; screening; mammography; ultrasound
MeSH Terms: conditions — Breast Neoplasms | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- group 1 (Experimental): screening with mammography alone
  Interventions: Other: mammography
- group 2 (Experimental): screening with ultrasonography alone
  Interventions: Other: ultrasound
- group 3 (Experimental): screening with both mammography and ultrasound
  Interventions: Other: mammography and ultrasound

INTERVENTIONS:
Other: mammography — participants were screened by mammography alone every year
  Arms: group 1
Other: ultrasound — participants were screened by ultrasound alone every year
  Arms: group 2
Other: mammography and ultrasound — Participants were screened by both mammography and ultrasound every year
  Arms: group 3

SUMMARY:
Early detection of breast cancer through screening has been a common practice in the United States and several European countries for decades.It is effective in reducing the mortality of breast cancer and improving the postoperative quality of life of patients. Mammography has been the standard imaging method for the screening, and in recent years, a supplemental ultrasound exam is also recommended.A prospective, multi-center, randomized trial is needed to define an optimal screening strategy that suits Chinese women and the socioeconomics of China.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent；
* residence from community or working units

Exclusion Criteria:

* pregnancy；
* lactation；
* known metastatic cancer；
* signs or symptoms of breast disease；
* presence of breast implants, breast surgery within prior 12 months；
* had mammography or ultrasound exam within prior 12 months
* males.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47709 (Actual)
Dates: Start 2008-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
screening yield | 3 years
  Sensitivities, specificities, positive predictive values, and negative predictive values

SECONDARY OUTCOMES:
Cost-effectiveness | 3 years
  cost of each screening modility to detect one cancer

CONTACTS AND LOCATIONS:
Overall Officials: Sun Qiang, MD, Study Chair — PUMCH
Locations (14):
- China (14):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing ChaoYang Hospital affiliated to the Capital Medical University, Beijing, Beijing Municipality
  - Beijing Hospital affiliated to Ministry of Health, Beijing, Beijing Municipality
  - Chinese 307 Hospital affiliated to the People's Liberation Army, Beijing, Beijing Municipality
  - First Hospital affiliated to Peking University, Beijing, Beijing Municipality
  - The Cancer Institute & Hospital, Peking Union Medical College Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - The General Hospital affiliated to Beijing Military Area Command, Beijing, Beijing Municipality
  - Southwest Hospital affiliated to the Third Military Medical University, Chongqing, Chongqing Municipality
  - Population and Family Planning Service Center of Zhuhai, Zhuhai, Guangdong
  - Maternity & Child Care Center of Qinhangdao, Qinhuangdao, Hebei
  - YingBin Surgery Hospital of Yancheng, Yancheng, Jiangsu
  - The Cancer Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - ShanXi Traditional Medicine Hospital, Taiyuan, Shanxi
  - The Cancer Hospital affiliated to Tianjin Medical University, Tianjin, Tianjin Municipality

REFERENCES:
- [Derived] Shen S, Zhou Y, Xu Y, Zhang B, Duan X, Huang R, Li B, Shi Y, Shao Z, Liao H, Jiang J, Shen N, Zhang J, Yu C, Jiang H, Li S, Han S, Ma J, Sun Q. A multi-centre randomised trial comparing ultrasound vs mammography for screening breast cancer in high-risk Chinese women. Br J Cancer. 2015 Mar 17;112(6):998-1004. doi: 10.1038/bjc.2015.33. PMID 25668012